CLINICAL TRIAL: NCT03924739
Title: A Nurse-coordinated Integrated Care Model to Support Decision-making and Self-care in Patients With Atrial Fibrillation: A Randomized Controlled Trial
Brief Title: A Nurse-coordinated Integrated Care Model for Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Polly Wai-Chi Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RGC14604418
Record Dates: First submitted 2019-04-16; First posted 2019-04-23 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Self-care; Model of care; Nurse-led; Disease management; Empowerment
MeSH Terms: conditions — Atrial Fibrillation; Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will participate in a 13-week, nurse-coordinated integrated care model.
  Interventions: Behavioral: Nurse-coordinated integrated care model for AF
- Control group (No Intervention): The control group will receive the conventional care provided by the study hospital.

INTERVENTIONS:
Behavioral: Nurse-coordinated integrated care model for AF — Participants in the intervention group will participate in a 13-week, nurse-coordinated integrated care model comprising the following care components intended to comprehensively address the needs of AF patients: 1) a risk profile assessment and shared decision-making regarding OAC use; 2) an empowerment-based educational module on AF self-care; 3) nurse-initiated telephone support; and 4) patient-initiated contact for professional advice.
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the effects of a nurse-coordinated, empowerment-based integrated care model on self-care behaviors and psychosocial outcomes in patients with atrial fibrillation (AF), and to explore how this intervention affects the self-care behaviors and quality of life from the patients' perspective.

Stroke prevention by oral anticoagulants (OAC) and control of arrhythmia and risk factors remain the cornerstones of AF management. However, under-prescription, non-adherence to treatment, and suboptimal anticoagulation control limit the efficacy of OACs. The poor abilities of patients regarding the self-control of arrhythmia and risk factors further contributes to worse outcomes. According to the World Health Organization, the best approach to chronic disease management involves the empowerment of patients to become active self-care agents. The literature indicates that a multifaceted, nurse-coordinated care model integrating all important care components with an empowerment approach could most effectively and actively engage patients in self-care.

This mixed-methods study comprises a randomized controlled trial and an exploratory qualitative study. A total of 392 community-dwelling patients aged ≥65 years with a confirmed diagnosis of AF, a high stroke risk, and no OAC treatment will be recruited from the medical outpatient clinics of a university-affiliated teaching hospital. The patients will be randomly allocated to intervention or control groups, which will receive treatment via the nurse-coordinated integrated care model or standard care, respectively. We hypothesize that compared to patients receiving standard care, AF patients exposed to the nurse-coordinated care model will be more likely to achieve compatible patient and physician decisions regarding the use of OAC, as well as better changes in medication adherence, anxiety, depression and health-related quality of life both immediately and 6 months post intervention.

This study will uniquely adopt an empowerment-based approach to equip patients as active agents in AF management through a nurse-coordinated integrated care model that comprehensively addresses their needs. The findings will advance our knowledge of patients' self-care behaviors in the context of AF and will provide a new model of care to improve health outcomes in this population.

DETAILED DESCRIPTION:
The proposed study will have two aims: i) to evaluate the effects of a nurse-coordinated integrated care model with a patient empowerment approach on the compatibility of patients' and physicians' decisions regarding oral anticoagulants (OAC) use, medication adherence, anxiety, depression, and health-related quality of life (HRQoL) and ii) to explore how and why the intervention affects health outcomes from the patients' perspectives. The first aim is based on a research hypothesis in which AF patients exposed to the nurse-coordinated integrated care model will be more likely to report achieving compatible patient and physician decisions regarding OAC use, better changes in medication adherence, anxiety, depression, and HRQoL, compared to patients who receive conventional care.

Study design This will be a sequential mixed-methods study with two phases. Phase 1 will comprise a prospective, single-blinded randomized controlled trial (RCT) to investigate the effects of the nurse-coordinated integrated care model on various health outcomes among patients with AF. Phase 2 will comprise an exploratory qualitative study to determine how and why the intervention works. After collecting baseline data, the research nurse (RA1) will randomly allocate patients into the intervention or control group. Block randomization (block size: 8, 10, or 12) will be used to ensure even participant distribution between the two groups. The block size and respective study group allocation sequence will be determined using a computer-generated sequence. Chronologically recruited patients will be allocated to the study groups by RA1 according to this computer-generated sequence. Participants allocated to receive the nurse-coordinated integrated care model will be provided with an appointment 1-2 weeks before their next scheduled medical appointment to initiate the intervention. The participants allocated to the control group will continue to receive conventional care as arranged by the hospital. An independent research assistant (RA2) who is blinded to the study group allocations will collect post-intervention data through medical record reviews and telephone interviews upon completion of the intervention and 6 months thereafter.

For Phase 2 of the study, a purposive sample of 30 participants from the intervention group will be invited to participate in a qualitative interview. Participants with different treatment responses to the nurse-coordinated integrated AF care model will be recruited according to changes in their post-intervention HRQoL scores. Ten participants will be selected from each range of HRQoL changes: 0-34th percentile, 35th-68th percentile, and >68th percentile.

Study interventions Intervention group: Nurse-coordinated integrated care model for AF Participants in the intervention group will participate in a 13-week, nurse-coordinated integrated care model comprising the following care components intended to comprehensively address the needs of AF patients: 1) a risk profile assessment and shared decision-making regarding OAC use; 2) an empowerment-based educational module on AF self-care; 3) nurse-initiated telephone support; and 4) patient-initiated contact for professional advice. The details of each care component of the intervention are described below.

1. Risk profile assessment and shared decision-making regarding OAC use A pre-consultation session will be provided 1-2 weeks before the patient's next medical clinic consultation. This session will comprise two components: an individualized assessment and a group-based session to enhance patients' participation in shared decision-making. First, RA1 will conduct a comprehensive, individualized risk assessment of patients. The risk assessment will address multiple aspects, including i) the stroke risk based on the CHA2DS2-VASc score, ii) bleeding risk based on the HAS-BLED score, and iii) quality of vitamin K antagonist (VKA) anticoagulation therapy based on the SAMe-TT2R2 score. Details of the CHA2DS2-VASc score were elaborated in a previous section of this proposal. The HAS-BLED score predicts the bleeding risk according to the following risk factors: hypertension, abnormal renal/liver function, stroke, bleeding history or predisposition, labile International normalized ratio (INR), age >65 years, and concomitant drug/alcohol use. The SAMe-TT2R2 score assesses the likelihood of poor INR control among patients with AF on VKA therapy according to sex, age, medical history, treatment, tobacco use, and race. These risk stratification scores provide information crucial to determining the optimal treatment options for each patient.

   After the risk assessment, the nurse will conduct a face-to-face session in a small-group (6-8 patients/group) format to empower patients regarding decision-making and communication with physicians. This face-to-face approach was selected in accordance with literature suggesting it to be more effective than a written format. Additionally, group teaching can promote peer learning and modeling. The session will begin with a structured educational session on AF and its complications, with emphasis placed on understanding the link between AF and ischemic stroke and the deleterious effects of rapid ventricular rates on cardiac function. The currently available and suitable OAC options (warfarin and Non-vitamin-K oral anticoagulants (NOACs)) and their pros and cons (including the self-financed nature of novel OAC) as well as the rationales for rate and rhythm control will also be discussed. To assist patients with decision-making regarding OAC use, a patient decision aid developed by the National Institute of Health and Care Excellence will be used. This aid organizes treatment options in an Option Grids format, wherein 10 frequently asked questions are presented vertically downwards with the options presented horizontally across the table. This format facilitates comparison and clarifies the options. Numeric and graphic formats with pictograms will be used to help patients understand the absolute and relative risks of a stroke when not using OACs or a major bleeding episode while using OACs. Patients' individual risk profiles will be used to illustrate their stroke risks with and without OAC and their bleeding risk with OAC in a graphical format. The nurse will present the risk and benefit information in a fair and balanced manner.

   Another care component will engage patients in shared decision-making regarding OAC use by empowering them to better communicate their decisions to physicians during upcoming medical consultations. This component will highlight the key points of assertive communication, including asking questions, expressing concerns, and stating opinions and preferences regarding OACs for stroke prevention. The patients will be encouraged to generate a list of questions and concerns to propose to their physicians. To enhance patients' confidence in their ability to maintain assertive communication in stressful situations, a series of scenario-based patient models in video format will be used to optimize the acquisition of skills for handling challenging encounters. A role-play-based rehearsal will be conducted to allow patients to practice their new skills and observe others' behavior. The nurse will debrief patients to discuss their performance and provide feedback. Throughout the session, the nurse will adopt a supportive and non-judgmental attitude.
2. Empowerment-based group educational module The same group of patients will attend an empowerment-based educational module beginning 1 week after their medical appointments. The module will comprise five weekly educational sessions covering the following major topics related to AF self-care: i) medication management, ii) symptom monitoring, iii) crisis management, iv) activities and exercise, and v) risk factor management to reduce risks of stroke and bleeding. The educational content of each session will comply with the recommendations of major practice guidelines for AF management.

   During each session, the nurse will implement the empowerment process to enhance patients' knowledge, skill acquisition, and confidence in AF self-care. The empowerment approach emphasizes the use of interactive teaching strategies, experiential learning, and self-reflection during the educational process to optimize learning. First, the nurse will deliver a structured educational session about the topic of the week. Emphasis will be placed on assisting patients with understanding the links between their self-care behaviors and health consequences to ensure that they appreciate the importance of their own efforts in managing AF. The nurse will encourage patients to share their current practices, and facilitate them to identify discrepancies between the suggested self-care and their current practices. The nurse will also highlight possible health consequences of these discrepancies and assist patients with setting self-directed goals related to those areas. After goal-setting, a subsequent interactive skill-building session will ensure that patients acquire the skills required to perform specific self-care behaviors. For example, to enhance patients' confidence regarding crisis management, a series of scenario-based patient models in video format will be used to optimize the acquisition of skills needed to handle challenging encounters related to possible crises, such as a major bleeding event or suspected stroke episode. A role-play-based rehearsal will be conducted, and the nurse will discuss the patients' performances and provide feedback. The nurse will make use of group dynamics by encouraging peer discussions of successful self-care actions, feelings, concerns, and perceived barriers to goal achievement. The nurse will also work with the patients to mutually develop action plans for achieving goals set during each weekly educational session. Each subsequent session will begin with a discussion of progress in goal attainment. Challenges and barriers faced while implementing the action plans set during the previous week will also be discussed.
3. Nurse-initiated telephone support The nurse will provide continued support by telephone after the face-to-face sessions have been completed (two weekly and two bi-weekly calls). A telephone record containing patients' clinical profiles, AF-related treatments, self-management goals, and action plans will be used to facilitate the process. The nurse will monitor patients' adherence, symptom profiles, treatment efficacies, adverse effects, and goal attainment progress; identify barriers in the self-care process; and provide resolutions and continued support via the telephone. Health counseling and advice given will be documented to guide subsequent telephone correspondence.
4. Patient-initiated contact for professional advice All participants from the intervention group will be provided with telephone access to the nurse for inquiries regarding disease management during office hours. The nurse will provide health advice and counseling accordingly. For severe undesirable symptoms and adverse reactions to medications, the nurse will attempt to advance patients' follow-up appointments or advise patients to seek emergency medical care if necessary. All correspondence and advice given will be documented in patients' profiles.

Control group: Conventional care The control group will receive the conventional care provided by the study hospital.

ELIGIBILITY:
Inclusion Criteria:

* age ≥65 years
* community-dwelling
* confirmed diagnosis of AF
* a CHA2DS2-VASc score of ≥1 in men and ≥2 in women
* no use of OAC therapy

Exclusion Criteria:

* impaired communication or cognitive abilities (i.e., an Abbreviated Mental Test score ≤6)
* or severe co-existing medical conditions (e.g., terminal illness) that would hinder participation in research activities

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 392 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) Questionnaire | Change from Baseline AFEQT at the 13th week (after the intervention) and 6 months (follow up)
  The 20-item AFEQT measures disease-specific HRQoL in AF patients using 4 subscales: symptoms, daily activities, treatment concerns, and treatment satisfaction. All subscales are rated on a 7-point Likert scale, with higher scores indicating a poorer HRQoL.

SECONDARY OUTCOMES:
Use of oral anticoagulants | At 6 months (follow up)
  A single item to assess whether the participants have been prescribed with an oral anticoagulant
Morisky, Green and Levine Adherence Scale (MGLS) | Change from Baseline MGLS at the 13th week (after the intervention) and 6 months (follow up)
  The 4-item MGLS will be used to assess self-reported medication adherence. Each item measures a specific medication-taking behavior using a dichotomous (yes/no) response. The wording of the questions was reversed to avoid 'yes-saying' bias. The sum of yes answers provides a composite measure of non-adherence.
Hospital Anxiety and Depression Scale (HADS) | Change from Baseline HADS at the 13th week (after the intervention) and 6 months (follow up)
  The 14-item Chinese-Cantonese version of the HADS will be used to measure anxiety and depression. This instrument is rated on a 4-point Likert scale, with higher scores indicating more intense anxiety and depression.
Decision concordance on oral anticoagulant between patients and physicians | At 6 months (follow up)
  A single item to evaluate whether patients and their attending physicians have the same decision on use of oral anticoagulants for stroke prevention

CONTACTS AND LOCATIONS:
Overall Officials: Polly Li, Dr, Principal Investigator — The University of Hong Kong, School of Nursing
Locations (1):
- The School of Nursing, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li PWC, Yu DSF, Yan BP. Nurse-led multi-component behavioural activation programme to improve health outcomes in patients with atrial fibrillation: a mixed-methods study and feasibility analysis. Eur J Cardiovasc Nurs. 2023 Sep 5;22(6):655-663. doi: 10.1093/eurjcn/zvac104. PMID 36394495
- [Derived] Li PWC, Yu DSF, Yan BBY. A nurse-coordinated integrated care model to support decision-making and self-care in patients with atrial fibrillation: A study protocol. J Adv Nurs. 2019 Dec;75(12):3749-3757. doi: 10.1111/jan.14164. Epub 2019 Aug 27. PMID 31350778

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT03924739/Prot_SAP_002.pdf
  • Informed Consent Form (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT03924739/ICF_001.pdf